CLINICAL TRIAL: NCT05397288
Title: Exercise Coaching Program With Aerobic Exercise and Resistance Exercise for Prefrail and Frail Older Adults
Brief Title: GrandMove Project to Promote Elders' Robustness Against Frailty
Acronym: GrandMove
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Simon K.Y.Lee Foundation (Unknown)
Responsible Party: Principal Investigator, Professor Terry Y.S. Lum, Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EA1511048
Record Dates: First submitted 2018-12-31; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Frail Elderly Syndrome
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance-Aerobic-Education (RAE) (Experimental): Participants first receive 6 months of resistance exercise, then 6 months of aerobic exercise, and finally 6 months of education program on healthy lifestyle.
  Behavioral: Resistance exercise (R) Behavioral: Aerobic exercise (A) Behavioral: Healthy lifestyle education (E)
  Interventions: Behavioral: Resistance exercise (R); Behavioral: Aerobic exercise (A); Behavioral: Healthy lifestyle education (E)
- Aerobic-Resistance-Education (ARE) (Experimental): Participants first receive 6 months of aerobic exercise, then 6 months of resistance exercise, and finally 6 months of education program on healthy lifestyle.
  Behavioral: Aerobic exercise (A) Behavioral: Resistance exercise (R) Behavioral: Healthy lifestyle education (E)
  Interventions: Behavioral: Resistance exercise (R); Behavioral: Aerobic exercise (A); Behavioral: Healthy lifestyle education (E)
- Education-Resistance-Aerobic (ERA) (Experimental): Participants first receive 6 months of education program on healthy lifestyle, then 6 months of resistance exercise, and finally 6 months of aerobic exercise.
  Behavioral: Healthy lifestyle education (E) Behavioral: Resistance exercise (R) Behavioral: Aerobic exercise (A)
  Interventions: Behavioral: Resistance exercise (R); Behavioral: Aerobic exercise (A); Behavioral: Healthy lifestyle education (E)

INTERVENTIONS:
Behavioral: Resistance exercise (R) — A 6-month program led by trained young-old exercise coaches consisting of structured training with 5 progressive levels of intensity, with protocols for implementation in a home surrounding and community center settings. During the 6-month program, group practice and home visit (individual) sessions (45 mins each) are delivered in a tapering schedule:
  * 1st month: group practice (1 time/week), home visits (2 times/week)
  * 2nd month: group practice (1 time/week), home visit (1 time/week), phone call (1 time/week)
  * 3rd month: group practice (1 time/week), phone calls (2 times/week)
  * 4th month: phone calls (2 times/week)
  * 5th month: phone calls (1 time/week)
  * 6th month: weaning period
Behavioral: Aerobic exercise (A) — A 6-month programs led by trained young-old exercise coaches consisting of structured training with 5 progressive levels of intensity, with protocols for implementation in a home surrounding and community center settings. During the 6-month program, group practice and home visit (individual) (45 mins each) are delivered in a tapering schedule:
  * 1st month: group practice (1 time/week), home visits (2 times/week)
  * 2nd month: group practice (1 time/week), home visit (1 time/week), phone call (1 time/week)
  * 3rd month: group practice (1 time/week), phone calls (2 times/week)
  * 4th month: phone calls (2 times/week)
  * 5th month: phone calls (1 time/week)
  * 6th month: weaning period
Behavioral: Healthy lifestyle education (E) — A 6-month program led by retired nurses covering topics including nutrition, sleep, medication, cognition, and exercising. During the 6-month program, group talks and individual consultation (45 mins each) are delivered in a tapering schedule:
  * 1st month: group talk (1 time/week), individual consultation (2 times/week)
  * 2nd month: group talk (1 time/week), individual consultation (1 time/week), phone call (1 time/week)
  * 3rd month: group talk (1 time/week), phone calls (2 times/week)
  * 4th month: phone calls (2 times/week)
  * 5th month: phone calls (1 time/week)
  * 6th month: weaning period

SUMMARY:
This is a single-blind, cluster randomized, cross-over trial to investigate the effectiveness of (1) a 6-month aerobic exercise program, (2) a 6-month resistance exercise program, versus (3) a 6-month psychoeducation program on healthy lifestyle for improving frailty, physical performance, and quality of life in frail/prefrail older persons. After 6 months, participants receive the other two programs in a pseudo random order to explore any effects of program sequence.

DETAILED DESCRIPTION:
This is a single-blind, cluster randomized, cross-over trial to investigate the effectiveness of (1) a 6-month aerobic exercise program led by trained young-old exercise coaches, (2) a 6-month resistance exercise program led by trained young-old exercise coaches, versus (3) a 6-month psychoeducation program on healthy lifestyle led by retired nurses for improving frailty, physical performance, and quality of life in frail/prefrail older persons. A total of 390 frail/prefrail older persons are randomized into one of the three programs in groups of 6 to 10 persons.

After 6 months, participants receive the other two programs in a pseudo random order to explore any effects of program sequence. The sequences are: (a) resistance exercise, aerobic exercise, psychoeducation; (b) aerobic exercise, resistance exercise, psychoeducation; and (c) psychoeducation, resistance exercise, aerobic exercise. The entire intervention period lasts for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* screened as frail or prefrail using cutoff scores of the 5-item FRAIL scale;
* living in the community and planned to reside in the area for the duration of the study;
* gave informed consent to participate in the study

Exclusion Criteria:

* heart failure, uncontrolled angina, severe pulmonary disease, or end-stage disease with a life expectancy of less than 18 months
* diagnosed dementia or a cutoff score falling below threshold suggestive of dementia using the clock-face test
* has another member of the household participating in the study
* difficulty in communication with study personnel due to speech or hearing problems
* other medical, psychiatric, or behavioural factors that may interfere with study participation or the ability to follow the intervention protocol

Temporary Exclusion Criteria:

* had stroke, hip fracture, myocardial infarction, major heart surgery, deep vein thrombosis, pulmonary embolus, spinal surgery, or hip or knee replacement within the previous 6 months;
* currently prescribed activity limitation or weight-bearing limitation by a formal healthcare professional;
* limited physical activity due to chest pain or dyspnoea without definitive treatment by a healthcare provider;
* currently consume more than 14 alcoholic drinks per week;
* currently enrolling in another randomized trial involving lifestyle or pharmacological interventions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 390 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change in physical frailty status measured by the 5-item FRAIL scale at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in physical frailty status is measured by the 5-item FRAIL scale at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 5, with 0 representing robust health status, 1-2 pre-frail, and 3-5 frail.
Change in physical performance measured by Short Physical Performance Battery (SPPB) at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in physical performance measured by Short Physical Performance Battery (SPPB) at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 12. Higher scores represent better physical performance, lower scores represent poor physical performance.
Change in upper body strength measured by 30-second bicep curl test at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in upper body strength measured by 30-second bicep curl test at baseline, 6 months, 12 months and 18 months. Performance is defined by the frequency of arm curls completed in 30 seconds while sitting in a chair. Higher frequencies represent better upper body strength, lower frequencies represent poor upper body strength.
Change in aerobic exercise capacity measured by 2-minute step test at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in aerobic exercise capacity measured by 2-minute step test at baseline, 6 months, 12 months and 18 months. Performance on the test is deﬁned as the number of right-side steps of the criterion height completed in 2 minutes. Higher frequencies represent better aerobic exercise capacity, lower frequencies represent poor aerobic exercise capacity.
Change in quality of life measured by World Health Organization Quality of Life - Older Adult Module (WHOQoL-OLD) at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in quality of life measured by World Health Organization Quality of Life - Older Adult Module (WHOQoL-OLD) at baseline, 6 months, 12 months and 18 months. It has a range of scores from 24 to 120. Higher scores indicate better quality of life, lower scores indicate poor quality of life.
Change in comprehensive frailty status measured by the 32-item Frailty Index (32-FI) at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in comprehensive frailty status measured by the 32-item Frailty Index (32-FI) at baseline, 6 months, 12 months and 18 months. The index is calculated by the sum score divided by the total number of valid responses, ranging from 0 to 1. Frailty status is defined as: robust (FI ≤ 0.08), prefrail (0.08 < FI < 0.25), and frail (FI ≥ 0.25).

SECONDARY OUTCOMES:
Change in handgrip strength measured by the (Jamar® Hand Dynamometer - Plus+ Digital - 200 lb. Capacity) at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in handgrip strength measured by the (Jamar® Hand Dynamometer - Plus+ Digital - 200 lb. Capacity) at baseline, 6 months, 12 months and 18 months. Performance is defined as the grip force exerted on the dynamometer. Larger forces indicate better handgrip strength, smaller forces indicate poor handgrip strength.
Change in pain severity measured by Face Pain Scale - Revised at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in pain severity measured by Face Pain Scale - Revised at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 10, with 0 representing no pain, 10 representing very much pain.
Change in physical activity measured by Physical Activity Scale for the Elderly (PASE) at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in physical activity measured by Physical Activity Scale for the Elderly (PASE) at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 361, with higher scores indicating higher physical activity level and lower scores indicating lower physical activity level.
Change in activities of daily living measured by Modified Barthel Index at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in activities of daily living measured by Modified Barthel Index at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 100, with higher scores indicating independence and lower scores indicating dependence.
Change in instrumental activities of daily living measured by Lawton Instrumental Activities of Daily Living at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in instrumental activities of daily living measured by Lawton Instrumental Activities of Daily Living at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 18, with higher scores indicating independence and lower scores indicating dependence.
Change in social network measured by Lubben Social Network Scale at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in social network measured by Lubben Social Network Scale at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 50 (scores <20 are classified as isolated; 21-25 as high risk for isolation; 26-30 as moderate risk for isolation; ≥ 31 as low risk for isolation).
Change in sleep quality measured by Pittsburgh Sleep Quality Index at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in sleep quality measured by Pittsburgh Sleep Quality Index at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 21, with higher scores indicating poor sleep quality and lower scores indicating better sleep quality.
Change in nutrition status measured by Mini Nutritional Assessment-Short Form at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in nutrition status measured by Mini Nutritional Assessment-Short Form at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 30 (scores of 24-30 are classified as normal nutritional status; 17-23.5 as at risk of malnutrition; <17 as malnourished).
Change in depressive symptoms measured by Patient Health Questionnaire - 9 (PHQ-9) at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in depressive symptoms measured by Patient Health Questionnaire - 9 (PHQ-9) at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression)
Change in extent of mobility measured by the Life Space Questionnaire at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in extent of mobility measured by the Life Space Questionnaire at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 9, reflecting the number of zones a person has moved in irrespective of the frequency and independence of these movements.
Change in verbal fluency was measured by the Verbal Fluency Test at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in verbal fluency was measured by the Verbal Fluency Test at baseline, 6 months, 12 months and 18 months. Performance is defined by the number of items in a category that can be verbally listed in 60 seconds. It has a range of scores from 0 to 20, with higher scores indicating higher verbal fluency and lower scores indicating lower verbal fluency.
Change in cognitive performance measured by Digit Symbol Substitution Test at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in cognitive performance measured by Digit Symbol Substitution Test at baseline, 6 months, 12 months and 18 months. Performance is defined by the number of correct symbols substitution in 90 seconds. It has a range of scores from 0 to 93, with higher scores indicating better cognitive performance and lower scores indicating poor cognitive performance.
Change in logical memory was measured by the Logical Memory Test at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in logical memory was measured by the Logical Memory Test at baseline, 6 months, 12 months and 18 months. Performance is defined as the number of correct word items recalled. It has a range of scores from 0 to 23, with higher scores indicating better logical memory and lower scores indicating poor logical memory.
Change in digit span measured by the Digit Span Test at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in digit span measured by the Digit Span Test at baseline, 6 months, 12 months and 18 months. The sequence and span scores have a range from 0 to 8 for forward subsets, and the sequence and span scores have a range from 0 to 7 for backward subsets. Higher scores indicating better cognitive performance and lower scores indicating poor cognitive performance.
Change in health literacy measured by Chinese Health Literacy for Chronic Care at baseline, 6 months, 12 months and 18 months. | 4 time points including: baseline, 6 months, 12 months, 18 months
  Change in health literacy measured by Chinese Health Literacy for Chronic Care at baseline, 6 months, 12 months and 18 months. It has a range of scores from 0 to 48, and the cut-off score is 36 (≥ 36 indicates "adequate health literacy").

OTHER OUTCOMES:
Change in body composition measured by Dual-energy X-ray absorptiometry (DEXA) scanning at baseline and 6 months (outcome in frail subgroup only). | 2 time points including: baseline, 6 months
  Change in body composition measured by Dual-energy X-ray absorptiometry (DEXA) scanning at baseline and 6 months (outcome in frail subgroup only). The test results will be in the form T score (a score of -1 or above is classified as normal; a score between -1.1 and -2.4 is classified as osteopenia (low bone mass); a score of -2.5 and below is defined as osteoporosis).
Change in functional muscular fitness measured by 30-second Chair Sit-to-stand Test at baseline and 6 months (outcome in frail subgroup only). | 2 time points including: baseline, 6 months
  Change in functional muscular fitness measured by 30-second Chair Sit-to-stand Test at baseline and 6 months (outcome in frail subgroup only). The score is the number of stands a person can complete in 30 seconds, with higher scores indicating better functional muscular fitness and lower scores indicating poor functional muscular fitness.
Change in upper and lower body strength measured by 3-repetition Maximum (3-RM) Test using Keiser pneumatic variable-resistance machines at baseline and 6 months (outcome in frail subgroup only). | 2 time points including: baseline, 6 months
  Change in upper and lower body strength measured by 3-repetition Maximum (3-RM) Test using Keiser pneumatic variable-resistance machines at baseline and 6 months (outcome in frail subgroup only). The score is defined as the maximum weight a person can lift for 3 repetitions.
Change in cardiovascular fitness measured by Ergometers and MedGrapics Ultima CardiO2 Gas Exchange System at baseline and 6 months (outcome in frail subgroup only). | 2 time points including: baseline, 6 months
  Change in cardiovascular fitness measured by Ergometers and MedGrapics Ultima CardiO2 Gas Exchange System at baseline and 6 months (outcome in frail subgroup only).
Change in balance measured by Multifunctional force-measuring plate at baseline and 6 months (outcome in frail subgroup only). | 2 time points including: baseline, 6 months
  Change in balance measured by Multifunctional force-measuring plate at baseline and 6 months (outcome in frail subgroup only).
Change in flexibility measured by Sit and Reach Flexibility Test at baseline and 6 months (outcome in frail subgroup only). | 2 time points including: baseline, 6 months
  Change in flexibility measured by Sit and Reach Flexibility Test at baseline and 6 months (outcome in frail subgroup only). The score is the recorded distance a person can reach forward by the hand with a seated position.

CONTACTS AND LOCATIONS:
Overall Officials: Terry YS Lum, PhD, Principal Investigator — HKU
Locations (1):
- The University of Hong Kong, Hong Kong, Non-US Or Canadian Address, Hong Kong

IPD SHARING:
Plan to Share IPD: No